CLINICAL TRIAL: NCT03012347
Title: Evaluation of a Gel Sunscreen in Controlled Use Conditions
Brief Title: Evaluation of a Gel Sunscreen in Controlled Use Conditions (208/2016)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19208
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunscreen Users (Experimental): Subjects will participate in a 2-Day study involving three applications of a single test article each day. The first application will be followed by an exposure of 30 minutes in a hot room.
  Interventions: Drug: BAY987517; Drug: BullFrog Gel Sunscreen Land Sport SPF-50

INTERVENTIONS:
Drug: BAY987517 — Subjects will be instructed to apply the test article in a split-body and face configuration, to the assigned side of the body (face, arms, torso, and legs), as they normally would before going outdoors for a run, walk or other sport related activity. (Formulation: RB# Y73-161)
Drug: BullFrog Gel Sunscreen Land Sport SPF-50 — Subjects will be instructed to apply the test article in a split-body and face configuration, to the assigned side of the body (face, arms, torso, and legs), as they normally would before going outdoors for a run, walk or other sport related activity.

SUMMARY:
To explore and quantify potential issues with application of a gel sunscreen in Outdoor Use testing, in a controlled indoor environment

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female.
* Subjects must be adults between 18 and 45 years of age.
* Subjects must have and have had a consistently active lifestyle for at least the previous few years (exercise
* outdoors and in direct sun exposure at least 2 times per week for at least 30 minutes-acceptable activities include tennis, running, jogging, walking, golf, etc.), i.e., outdoor activity should not be a new behavior.
* Subjects must have used a sunscreen with SPF 50 or higher within the previous 9 months.

Exclusion Criteria:

* Subjects who have received or used an Investigational New Drug within the last 30 days.
* Subjects who have been active participants in another clinical or subjective product performance study within the last 30 days.
* Subjects who have a known allergy or sensitivity to sunscreen ingredients or test materials.
* Subjects with respiratory allergies or asthma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Feeling any discomfort after applying the product assessed by questionnaire | 15 minutes after each application

CONTACTS AND LOCATIONS:
Locations (1):
- Memphis, Tennessee, United States